CLINICAL TRIAL: NCT05398211
Title: Music Therapy as a Treatment for Delirium in Acutely Hospitalized Older Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Academy of Music (Other); University of Melbourne (Other)
Responsible Party: Principal Investigator, Bjørn Erik Neerland, MD, Principal Investigator, MD, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REK 457017
Record Dates: First submitted 2022-05-13; First posted 2022-05-31 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Delirium in Old Age; Delirium of Mixed Origin; Delirium Superimposed on Dementia; Delirium Confusional State
Keywords: music interventions; music therapy; delirium; acute confusion; treatment; severity; acute geriatrics; arousal; attention; cognition
MeSH Terms: conditions — Delirium; Confusion

STUDY DESIGN:
Intervention Model Description: A randomized controlled repeated measures design.
Who Masked: Outcomes Assessor
Masking Description: Masking of the therapist and the participants will not be possible, due to the nature of the interventions. Additionally, the music therapist will need to be acquainted with the results of the randomization in order to tailor each individual intervention. Masking of the outcome assessors will be attempted, but is expected to be incomplete, since the assessors will have to related to both the patients directly and to the medical staff who are well-acquainted with the patients, and who both might accidentally reveal the treatment allocation. Outcome assessors will attempt to remind the medical staff to keep the allocation concealed at all times. In order to verify the masking, the assessors will be asked about their knowledge of the patients' allocation to the treatment groups upon the last completed assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preferred Recorded Music (PRM) (Experimental): The Preferred Live Music (PLM) aims to elicit participants' responses from live music and the ensuing musical and non-musical interactions with the music therapist (MT). In the PLM intervention, preferred songs performed live on guitar or electronic keyboard will be played by a credentialed MT. When appropriate participants may also play percussion instruments offered to them. Elements of improvisation will be incorporated to allow for active engagement by the participants, and to provide opportunities for musical and non-musical attunement to emerge.
  Interventions: Behavioral: Preferred Recorded Music (PRM)
- Preferred Live Music (PLM) (Experimental): The Preferred Recorded Music (PRM) intervention aims to detect responses directly attributable to the music. Participants listen to pre-recorded preferred originally-published versions of music accessed by Spotify music-streaming service and played through loud-speakers. The MT will only start the music, and otherwise not be present during the interventions to ensure the minimal direct interaction with the participants.
  Interventions: Behavioral: Preferred Live Music (PLM)

INTERVENTIONS:
Behavioral: Preferred Recorded Music (PRM) — Preferred Recorded Music (PRM) involves a credentialed music therapist in planning and administering, which qualifies it as music therapy, which is defined as a professional use of music and its elements to improve physical, social, communicative, emotional, intellectual, and spiritual health, optimize quality of life and wellbeing(Aigen, 2013; Bruscia, 2014). PRM intervention will be delivered for 30 minutes, once per day at the same time of the day, for three consecutive days. The intervention will consist of the previously assessed preferred songs/musical pieces. During the PRM intervention the MT will start/stop the music and otherwise not engage with the participants during the listening session.
  Arms: Preferred Recorded Music (PRM)
Behavioral: Preferred Live Music (PLM) — Preferred Live Music (PLM) involves a credentialed music therapist in planning and administering which qualifies it as music therapy, which is defined as professional use of music and its elements to improve physical, social, communicative, emotional, intellectual and spiritual health, optimize quality of life and wellbeing (Aigen, 2013; Bruscia, 2014).PRM intervention will be delivered for 30 minutes, once per day at the same time of the day, for three consecutive days. The intervention will consist of the previously assessed preferred songs/musical pieces. The MT will be more actively engaged in a musical interaction with the participants in the PLM interventions.
  Arms: Preferred Live Music (PLM)

SUMMARY:
The purpose of this study is to assess feasibility and potential effectiveness of two different music interventions for managing delirium symptoms in acute geriatric patients.

DETAILED DESCRIPTION:
Delirium is a neuropsychiatric syndrome characterized by an acute alteration in attention, awareness, arousal and cognition, precipitated by an acute illness, intoxication, trauma or surgery. It is highly prevalent in older, frail and acutely hospitalized patients, and associated with poor outcomes, with few effective treatment alternatives. Non-pharmacological interventions and music show promising effects.

This study protocol aims to determine whether music interventions (MIs) delivered by a credentialed music therapist, are feasible and effective for regulating delirium symptoms in acute geriatric patients and whether the standardized delirium tools are sensitive to detect observable responses. Primary, feasibility outcomes are evaluating recruitment rate, treatment fidelity and adherence, as well as feasibility and accuracy in data collection procedures. Main effect-outcome is delirium severity, but delirium duration, cognitive status, length of hospital stay, and medication use will also be recorded. The randomised repeated measures controlled trial design will record the participant responses before and after exposure to MIs (+/- 2 hours). Participants with delirium from an acute geriatric ward will be randomized to either live or recorded MI. Each intervention will be delivered to n=30 participants (n=60 in total), for 30 minutes, over three consecutive days. Ethical approval has been obtained from Regional Ethics Committee South East Norway.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 65 and with delirium or possible delirium at admission or detected within the last 72 hours, and still present.
* Appropriate informed consent is obtained.
* Participants will not be excluded if they are under long term care and have comorbidities such as dementia or mild cognitive impairment.
* Patients will not be excluded if they have Covid-19.

Exclusion Criteria:

* Patients who were previously enrolled, and were readmitted during the study period will not be re-included.
* The patients with severe hearing impairments, severe psychiatric conditions, and/or severe alcohol/substance addiction where that is the main reason for admission will be excluded.
* The patients whose assessed musical preferences involve orchestral or other kinds of music which cannot be performed live by voice and a guitar.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Up to 52 weeks
  How many participants were recruited and randomized per month on average from those eligible, calculated by dividing the total number of the participants recruited by the total number of months that the trial recruited for.
Retention and attrition rates | Up to 52 weeks
  Retention is defined as trial completion on study intervention, and will be calculated by dividing the number of participants completing the study by the total number of participants recruited. Attrition rates will be estimated by the percentage of participants that withdrew from the study, and calculated by dividing the number of the participants who withdrew by the total number recruited.
Adherence and deviations rates | Up to 52 weeks
  Adherence to the study protocol is defined as compliance with the described study protocol, and protocol deviations as any change or divergence from the study protocol for each participant. Adherence rate will be estimated by calculating the percentage of the music sessions (interventions) actually completed from those described in the protocol (by dividing the number of completed sessions by the number of planned sessions), and deviation rates will be measured by counting the deviations per participant during their participation in the study.
Treatment fidelity rating and internal and external validity of the study | Up to 52 weeks
  The level of treatment fidelity will be determined using NIH Behavioral Change Consortium questionnaire which assesses 5 mutually exclusive categories: study design, training, delivery, receipt, and enactment. The tool lists 25 fidelity attributes that should be rated dichotomously as:" Present", "Absent but should be present", or "Not applicable".

SECONDARY OUTCOMES:
Delirium severity | Up to 7 days
  Delirium severity as assessed by Observational Scale of Level of Arousal (OSLA), Richmond Agitation Sedation Scale (RASS).
Cognitive status | Up to 7 days.
  Pre-post interventions changes in attention, orientation and short-term memory, assessed by backwards tests and digit span tests, recall tasks and orientation questions from Memorial Delirium Assessment Scale-MDAS)
Duration of delirium during hospital stay | Up to 3 weeks.
  As diagnosed according to Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) criteria
Use of "rescue medication" during hospital stay | Up to 3 weeks.
  The total number of psycho-pharmacological medications per patients will be registered.
Length of hospital stay | Up to 3 weeks.
  The total number of days from admittance to the Acute Geriatric Department to discharge from hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Golubovic J, Neerland BE, Simpson MR, Johansson K, Baker FA. A randomized pilot and feasibility trial of live and recorded music interventions for management of delirium symptoms in acute geriatric patients. BMC Geriatr. 2025 May 2;25(1):306. doi: 10.1186/s12877-025-05954-1. PMID 40316916